CLINICAL TRIAL: NCT07231861
Title: An Open-Label, Randomized, Fasting, Single-Dose, Two-Sequence, Two-Period Crossover Study to Evaluate the Bioequivalence of "AJU-R713" and "R713R" in Healthy Adult Volunteers
Brief Title: Bioequivalence Study of AJU-R713 and R713R in Healthy Adult Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 25BA11701
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Bronchial Asthma; Perennial Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranlukast Test Formulation (Experimental): Two-period, single-dose, crossover study
  Interventions: Drug: AJU-R713; Drug: R713R
- Pranlukast Reference Formulation (Experimental): Two-period, single-dose, crossover study (reversed order)
  Interventions: Drug: AJU-R713; Drug: R713R

INTERVENTIONS:
Drug: AJU-R713 — Oral formulation
Drug: R713R — Oral formulation

SUMMARY:
To Evaluate the Safety and Pharmacokinetics of Pranlukast hydrate in Healthy Adults.

DETAILED DESCRIPTION:
This study evaluates the pharmacokinetic characteristics and safety of pranlukast in healthy adults. It is a randomized, open-label, single-dose, two-period crossover trial conducted under fasting conditions. Pharmacokinetic samples are collected up to 24 hours after dosing, and standard safety assessments are performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 years or older at the time of screening.
* Body mass index (BMI) between 18 and 30 kg/m².

  * Male subjects: body weight ≥ 50 kg.
  * Female subjects: body weight ≥ 45 kg.
* Clinically healthy based on medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory test results, as determined by the investigator.
* Willing and able to provide written informed consent after receiving a full explanation of the study.
* Subjects (and their partners, if applicable) agree to use highly effective, non-hormonal contraception from the first dosing day until one week after the last dose.

Exclusion Criteria:

* Use of drugs known to induce or inhibit drug-metabolizing enzymes within 30 days prior to the first dose, or any medication likely to interfere with the study within 10 days prior to dosing.
* Participation in any clinical trial involving investigational products within 6 months prior to the first dose.
* Whole blood donation within 8 weeks, or component blood donation within 2 weeks prior to the first dose.
* History of gastrointestinal surgery that may affect drug absorption (excluding appendectomy and hernia repair).
* Known hypersensitivity to the investigational product or its components.
* Known metabolic or genetic disorders such as galactose intolerance, lactase deficiency, glucose-galactose malabsorption, or phenylketonuria.
* History of clinically significant psychiatric illness.
* Pregnant or breastfeeding women, or women with a possibility of pregnancy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cmax of Pranlukast | 0 hour ~ 24 hour after drug administration
  To assess the maximum observed plasma concentration (Cmax) of Pranlukast
AUCt of Pranlukast | 0 hour ~ 24 hour after drug administration
  To assess the plasma concentration-time curve from time 0 to the last measurable concentration (AUCt) of Pranlukast

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea